CLINICAL TRIAL: NCT05722314
Title: ENDOMED: Evaluation of the Evolution of Endometriosis Lesions on MRI Before and After Medical Treatment.
Brief Title: ENDOMED: Evaluation of the Evolution of Endometriosis Lesions on Imaging Under Medical Treatment
Acronym: ENDOMED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOMED FIGUIER
Record Dates: First submitted 2022-12-22; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-11

CONDITIONS: Endometriosis Pelvic
Keywords: Endometriosis; hormonal treatment; Endometrioma; MRI; Deep Endometriosis; rectovaginal nodule
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometriosis is a difficult disease to diagnose because the symptoms are varied, unspecific and inconsistent from one patient to another. Magnetic resonance imaging is the gold standard for the diagnosis, staging and follow-up of this pathology. Moreover, the management of endometriosis can be medical or surgical depending on the severity and location of the lesions and the patient's expectations. The recommendations of the National College of Obstetricians and Gynecologists and the French National Health Authority are medical treatment first in a certain number of situations. These patients undergoing medical treatment then require close clinical and radiological follow-up in order to evaluate the effectiveness of the treatment and the evolution of the disease. The literature describes the appearance of endometriosis lesions on pelvic MRI quite well for the establishment of the diagnosis, but there are few data on the evolution and imaging description of these lesions when hormonal treatment is in progress. Thus, we decided to evaluate and describe the evolution of endometriosis lesions on magnetic resonance imaging under medical treatment and to examine a correlation between this radiological evolution and the clinical evolution of the patients.

DETAILED DESCRIPTION:
D-0 Consultation: The patient is referred to one of the gynecologists in our department to assess a suspected endometriosis.

If the symptomatology is suggestive of endometriosis and the patient has not yet had an MRI, it will be performed in the department. In all cases, the inclusion MRI will be performed or reviewed by the department's referring radiologists.

The patient is then offered to participate in the NoEndo (national observatory of endometriosis) project. Via this application, the patient will be able to fill in questionnaires evaluating her quality of life and pain (SF 36, EHP 30, EHP 5, FSFI, GIQLI).

In addition, the patient's history, age, BMI, type and duration of treatment and clinical examination will be collected via the NoEndo application. The initial therapeutic choice between hormonal treatment (with details of the choice of the molecule and dosage) or first management in MAP (medical assistance for procreation) (with details of the therapeutic sequence chosen) or therapeutic abstention (with details of the reason) will be collected in the NoEndo application.

M-6 Consultation: At 6 months of treatment, the patient will be seen in consultation, to assess her tolerance to the treatment undertaken. She will be asked to fill in the questionnaires evaluating her quality of life and pain. Any change in treatment or therapeutic strategy will be notified.

Patient compliance and whether or not amenorrhea was achieved will be recorded. M-12 MRI: At 12 months, the patient will have a new MRI check-up in our reference center at the CHU of Clermont-Ferrand according to the same modalities as the first examination and according to the service protocol.

M-12 Consultation: We will see the patient again in consultation, to evaluate again her tolerance of the treatment as well as her compliance. We will evaluate her pain as well as the results of the quality of life questionnaires that she will have filled out beforehand via the NoEndo application. We will also analyze the results of the MRI.

We will then discuss with the patient the various possible management options for the future: continuation of medical treatment, PMA course, surgery.

If the patient is or has been pregnant before the one-year MRI, the information will be notified and the surveillance MRI may be delayed.

ELIGIBILITY:
Inclusion Criteria:

* No history of endometriosis surgery
* Diagnosis of endometriosis suspected by an MRI performed or reviewed in a reference center
* Presence of symptomatology requiring medical treatment

Exclusion Criteria:

* Pregnant or postmenopausal patient
* Not speaking French, not affiliated to the french social security system
* Minors or under guardianship
* Need for surgical management in the first instance
* Contraindication to MRI (claustrophobia, renal insufficiency, gadolinium allergy, intracorporeal presence of metallic implant)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: Patients whose MRI results are in favor of deep endometriosis, taking medical treatment or included in a MAP program or in whom it is agreed to withhold treatment (by patient choice, refusal of initial medical or surgical management, desire for spontaneous pregnancy, etc.).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of lesions | 2 years
  To compare endometriosis lesions on pelvic MRI before and after one year of hormonal treatment. The size, appearance and location of the lesions will be compared

SECONDARY OUTCOMES:
Clinical evaluation | 2 years
  Evaluate the clinical evolution of patients undergoing medical treatment, based on the evolution of the Medical Outcomes Study Short Form (MOS SF-36) score, generalist quality of life questionnaire used in endometriosis
Clinical evaluation 2 | 2 years
  Evaluate the clinical evolution of patients undergoing medical treatment, based on the evolution of the Endometriosis Health Profile 30 (EHP-30) score, quality of life questionnaire specialized for endometriosis.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Figuier, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No